CLINICAL TRIAL: NCT02877368
Title: Sarcopenia in Patients With Gastrointestinal Stromal Tumours
Acronym: SARCO-GIST
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao003
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Gastrointestinal Stromal Tumours
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- gastrointestinal stromal tumours: Patients with advanced or high-risk resected gastrointestinal stromal tumours (GIST) .
  Interventions: Other: Computed tomography

INTERVENTIONS:
Other: Computed tomography

SUMMARY:
The treatment of advanced gastrointestinal stromal tumours (GIST) has shifted since the arrival of targeted therapies. Imatinib is an active multikinase inhibitor that mainly targets C-kit tyrosine-kinase receptors and the platelet-derived growth factor receptor. Imatinib use has been validated for adjuvant and palliative therapy settings. Imatinib is generally well-tolerated and known to improve performance status but up to 16% grades 3-4 toxicities, leading to at least 40% withdrawals, have been reported.

Recently, in oncology, sarcopenia was shown to be a predictor of severe toxicity patients included in phase 1 trials, suggesting that it should be considered an inclusion criterion for such studies. Sarcopenic patients had low performance status, shorter survival, more chemotherapy toxicities and post-operative infections, and longer post-operative hospitalization times. In addition, exposure to tyrosine-kinase inhibitors (e.g. sorafenib or sunitinib) has been associated with dose-limiting toxicity (DLT) in patients with renal cell or hepatocellular carcinomas.

Computed tomography (CT) scans acquired during routine care have been validated as an accurate and robust imaging technique to evaluate sarcopenia in cancer patients.

DETAILED DESCRIPTION:
Aims of the study were:

* to assess the influence of imatinib on sarcopenia patients with advanced or high-risk resected gastrointestinal stromal tumours (GIST)
* to compare imatinib-induced toxicities between patients with advanced or high-risk resected gastrointestinal stromal tumours (GIST) with pre-treatment sarcopenia and patients with advanced or high-risk resected gastrointestinal stromal tumours (GIST) without pre-treatment sarcopenia

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or high-risk resected gastrointestinal stromal tumours (GIST)
* Patients treated with imatinib prescribed at a fixed dose of 400 mg/day from 1 January 2005 to 31 December 2013
* Aged > 18 years

Exclusion Criteria:

* Patients who did not have CT imaging within the 30 days preceding treatment onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or high-risk resected gastrointestinal stromal tumours (GIST) with imatinib prescribed at a fixed dose of 400 mg/day.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
sarcopenia | Day 0
  Sarcopenia was defined for men by lumbar skeletal muscle index <53 cm2/m2 with body mass index >25 kg/m2 and <43 cm2/m2 with body mass index <25 kg/m2 Sarcopenia was defined for women, by lumbar skeletal muscle index <41 cm2/m2 with any body mass index.

SECONDARY OUTCOMES:
Imatinib-induced toxicities | Month 3
  Toxicity regarding all site (cutaneous with edema, rash, pruritus, xerosis, digestif with nausea, diarrhea, vomiting, biology with anemia, neutropenia, hepatitis,general with asthenia, muscle cramps musculaires, arthralgia), graded according to the National Cancer Institute Common Toxicity Criteria, version 3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Moryoussef F, Dhooge M, Volet J, Barbe C, Brezault C, Hoeffel C, Coriat R, Bouche O. Reversible sarcopenia in patients with gastrointestinal stromal tumor treated with imatinib. J Cachexia Sarcopenia Muscle. 2015 Dec;6(4):343-50. doi: 10.1002/jcsm.12047. Epub 2015 Jun 4. PMID 26673372